CLINICAL TRIAL: NCT00552929
Title: A Multi -Center, Randomized, Open -Label, Prospective Bridging, Parallel Dose-Finding Trial Comparing Efficacy, Safety and Pharmacokinetics of 5 Doses of Org 25969 Administered at 1-2 PTC After Rocuronium or Vecuronium in Japanese and Caucasian Subjects. Part B: Caucasian Subjects.
Brief Title: A Bridging Trial Comparing Sugammadex (Org 25969) at 1-2 Post-Tetanic Count (PTC) in Caucasian Participants. Part B (P05974)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05974; 2005-001133-15 (EudraCT Number); MK-8616-036 (Other: Merck Protocol Number); P05974 (Other: Schering-Plough Protocol Number); 19.4.209B (Other: Organon Protocol Number)
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Sugammadex 0.5 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered intravenously (IV), followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the second twitch (T2) response to Train-of-four (TOF) stimulation, a single dose of 0.5 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 1.0 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 1.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 2.0 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 2.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 4.0 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 4.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 8.0 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 8.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 0.5 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 0.5 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 1.0 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 1.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 2.0 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 2.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 4.0 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 4.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 8.0 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.03 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 8.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — After induction of anesthesia an intubation dose of a neuromuscular blocking agent (NMBA) was administered IV: either 0.9 mg/kg rocuronium (arms 1-5) or 0.1 mg/kg vecuronium (arms 6-10). Maintenance doses of 0.1-0.2 mg/kg rocuronium IV or 0.02-0.03 mg/kg vecuronium IV could be administered if necessary.
  At reappearance of T2 the randomized single dose of sugammadex (0.5 to 8.0 mg/kg) IV was administered.
  Other Names: Org 25969; MK-8616; Bridion^TM

SUMMARY:
The objective of the trial was to establish the dose-response relation of sugammadex given as a reversal agent of rocuronium or vecuronium at 1-2 Post-Tetanic Count (PTC) during sevoflurane anesthesia for Caucasian participants

ELIGIBILITY:
Inclusion Criteria:

* Participants of American Society of Anesthesiologists (ASA) class 1 - 3;
* Participants at least 20 years but under 65 years of age;
* Caucasian participants ;
* Participants scheduled for elective surgery requiring muscle relaxation in supine position and under sevoflurane anesthesia, in need of administration of a neuromuscular blocking agent (NMBA), with an anticipated duration of about 1.5- 3 hours;
* Participants who had given written informed consent. This was obtained before the investigator or the sub-investigator performed any procedures or assessments for the screening, and after the participant was informed about the nature and purpose of the study, the study procedures, and the risks and restrictions of the study.

Exclusion criteria:

* Participants in whom a difficult intubation because of anatomical malformations was expected;
* Participants known or suspected to have neuromuscular disorders impairing neuromuscular blockade (NMB) and/or significant renal dysfunction (for example a creatinine level > 1.6 mg/dl) and/or severe hepatic dysfunction.
* Participants known or suspected to have a (family) history of malignant hyperthermia;
* Participants known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia;
* Participants receiving medication expected to interfere with the rocuronium or vecuronium given in this trial, based on the dose and time of administration;
* Female participants who were pregnant;
* Female participants of childbearing potential not using birth control or using only oral contraception as birth control;
* Participants who were breast-feeding;
* Participants who had already participated in CT 19.4.209B, or in another trial with sugammadex;
* Participants who had participated in another clinical trial, not preapproved by Organon, within 6 months of entering into CT 19.4.209B.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2005-10-04 (Actual); Primary Completion 2006-09-15 (Actual); Study Completion 2006-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Duvaldestin P, Kuizenga K, Saldien V, Claudius C, Servin F, Klein J, Debaene B, Heeringa M. A randomized, dose-response study of sugammadex given for the reversal of deep rocuronium- or vecuronium-induced neuromuscular blockade under sevoflurane anesthesia. Anesth Analg. 2010 Jan 1;110(1):74-82. doi: 10.1213/ANE.0b013e3181c3be3c. Epub 2009 Nov 21. PMID 19933538
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in seven centers in Europe: one center in Belgium, one center in Denmark, three centers in France, and two centers in The Netherlands.
Groups:
- Sugammadex 0.5 mg/kg (Rocuronium): Sugammadex 0.5 mg/kg administered as a single-bolus intravenous (IV) dose at 1-2 posttetanic count (PTC) after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 1.0 mg/kg (Rocuronium): Sugammadex 1.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 2.0 mg/kg (Rocuronium): Sugammadex 2.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 4.0 mg/kg (Rocuronium): Sugammadex 4.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 8.0 mg/kg (Rocuronium): Sugammadex 8.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 0.5 mg/kg (Vecuronium): Sugammadex 0.5 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.3 mg/kg if necessary.
- Sugammadex 1.0 mg/kg (Vecuronium): Sugammadex 1.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.3 mg/kg if necessary
- Sugammadex 2.0 mg/kg (Vecuronium): Sugammadex 2.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.3 mg/kg if necessary
- Sugammadex 4.0 mg/kg (Vecuronium): Sugammadex 4.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.3 mg/kg if necessary
- Sugammadex 8.0 mg/kg (Vecuronium): Sugammadex 8.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.3 mg/kg if necessary
Period: Overall Study
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuronium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
Started (Randomized Participants) | 9 | 10 | 10 | 11 | 10 | 10 | 10 | 11 | 10 | 11
Participants as Treated | 9 (One participant randomized to sugammadex 0.5 mg/kg received sugammadex 3.7 mg/kg (4.0 mg\kg group)) | 10 | 10 | 11 (One participant randomized to sugammadex 0.5 mg/kg received sugammadex 3.7 mg/kg (4.0 mg\kg group)) | 10 | 9 | 10 | 11 | 10 | 11
Completed | 9 | 10 | 10 | 11 | 10 | 9 | 10 | 11 | 9 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Not Eligible | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall Number of Participants Receiving Sugammadex + Rocuronium or Sugammadex + Vecuronium as treated
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuronium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium) | Total
Number analyzed (Participants) | 9 | 10 | 10 | 11 | 10 | 9 | 10 | 11 | 10 | 11 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (7) | 42 (9) | 49 (6) | 51 (13) | 52 (9) | 44 (14) | 50 (14) | 54 (6) | 40 (11) | 50 (9) | 48 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 6 | 5 | 4 | 6 | 4 | 3 | 5 | 44
  Male | 5 | 8 | 5 | 5 | 5 | 5 | 4 | 7 | 7 | 6 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 9 | 9 | 10 | 11 | 10 | 9 | 9 | 11 | 10 | 11 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
American Society of Anaesthesiologists (ASA) Class [Count of Participants; unit: Participants] — ASA class Classification of physical status:
  ASA class 1: A normal healthy participant; ASA class 2: A participant with a mild systemic disease; ASA class 3: A participant with a severe systemic disease that limits activity, but is not incapacitating; ASA class 4: A participant with an incapacitating systemic disease that is a constant threat to life; ASA class 5: A moribund participant not expected to survive 24 hours with or without operation
  Participants
    ASA Class 1 | 6 | 5 | 2 | 6 | 5 | 7 | 8 | 7 | 9 | 6 | 61
    ASA Class 2 | 3 | 5 | 7 | 5 | 5 | 2 | 2 | 4 | 1 | 5 | 39
    ASA Class 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Sugammadex Administration to Recovery of the Neuromuscular Response to a Ratio of 0.9 for Train-Of-Four (TOF) Stimulation
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from neuromuscular blockade (NMB). In this study, twitch responses were recorded until the T4/T1 Ratio reached >= 0.9, the minimum acceptable ratio that indicated recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.9 indicates a faster recovery from NMB.
Time Frame: Up to 131:40 (min:sec)
Population: The analysis population consisted of all randomized and treated participants who had at least one post-baseline efficacy measurement, without any major or multiple minor protocol violations.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Sugammadex 1.0 mg/kg (Rocuroniium): Sugammadex 1.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuroniium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
Number analyzed (Participants) | 8 | 9 | 10 | 10 | 10 | 7 | 9 | 11 | 8 | 10
Minutes | 79.78 (33.02) | 28.00 (43.73) | 3.17 (1.52) | 1.65 (0.65) | 1.13 (0.33) | 68.40 (31.93) | 25.12 (24.87) | 9.08 (20.55) | 3.30 (3.45) | 1.65 (0.75)

2. Secondary Outcome: Time From Start of Sugammadex Administration to a T4/T1 Recovery Ratio of 0.7
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.7 indicates a faster recovery from NMB.
Time Frame: Up to 96:24 (min:sec)
Population: The analysis population consisted of all randomized and treated participants who had at least one post-baseline efficacy measurement, without any major protocol violation.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuroniium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
Number analyzed (Participants) | 8 | 10 | 10 | 10 | 10 | 8 | 9 | 11 | 9 | 10
Minutes | 47.72 (27.62) | 4.47 (1.95) | 2.17 (0.97) | 1.25 (0.52) | 0.93 (0.25) | 30.22 (34.70) | 4.07 (2.02) | 2.32 (1.20) | 1.65 (0.67) | 1.33 (0.57)

3. Secondary Outcome: Time From Start of Sugammadex Administration to a T4/T1 Recovery Ratio of 0.8
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.8 indicates a faster recovery from NMB.
Time Frame: Up to 102:25 (min:sec)
Population: The analysis population consisted of all randomized participants who were given at least one administration of sugammadex and had at least one post-baseline efficacy measurement, without any major protocol violation.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuroniium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
Number analyzed (Participants) | 8 | 10 | 10 | 10 | 10 | 7 | 9 | 11 | 9 | 10
Minutes | 57.00 (32.97) | 14.22 (20.62) | 2.45 (1.12) | 1.35 (0.57) | 0.98 (0.32) | 45.93 (29.55) | 5.10 (2.70) | 2.92 (1.75) | 2.87 (3.25) | 1.43 (0.58)

4. Secondary Outcome: Number of Participants With An Adverse Event (AE)
Description: The number of participants who had at least one AE during treatment and follow-up was assessed. An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: From Screening to 7 post-operative days
Population: All randomized participants who received at least one dose of study treatment and had follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuroniium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
Number analyzed (Participants) | 9 | 10 | 10 | 11 | 10 | 9 | 10 | 11 | 10 | 11
Participants | 6 | 8 | 8 | 10 | 8 | 6 | 6 | 7 | 6 | 8

ADVERSE EVENTS:
Time Frame: Up to 7 post-operative days
Description: All randomized participants who received at least one dose of study treatment and had follow-up.
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuronium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/10 | 0/11 | 0/10 | 0/9 | 0/10 | 0/11 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/10 | 1/10 | 1/11 | 0/10 | 0/9 | 0/10 | 0/11 | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 6/9 | 8/10 | 8/10 | 10/11 | 8/10 | 6/9 | 6/10 | 7/11 | 6/10 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 0.5 mg/kg (Rocuronium) (N=9) | Sugammadex 1.0 mg/kg (Rocuronium) (N=10) | Sugammadex 2.0 mg/kg (Rocuronium) (N=10) | Sugammadex 4.0 mg/kg (Rocuronium) (N=11) | Sugammadex 8.0 mg/kg (Rocuronium) (N=10) | Sugammadex 0.5 mg/kg (Vecuronium) (N=9) | Sugammadex 1.0 mg/kg (Vecuronium) (N=10) | Sugammadex 2.0 mg/kg (Vecuronium) (N=11) | Sugammadex 4.0 mg/kg (Vecuronium) (N=10) | Sugammadex 8.0 mg/kg (Vecuronium) (N=11)
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Vascular disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sugammadex 0.5 mg/kg (Rocuronium) (N=9) | Sugammadex 1.0 mg/kg (Rocuronium) (N=10) | Sugammadex 2.0 mg/kg (Rocuronium) (N=10) | Sugammadex 4.0 mg/kg (Rocuronium) (N=11) | Sugammadex 8.0 mg/kg (Rocuronium) (N=10) | Sugammadex 0.5 mg/kg (Vecuronium) (N=9) | Sugammadex 1.0 mg/kg (Vecuronium) (N=10) | Sugammadex 2.0 mg/kg (Vecuronium) (N=11) | Sugammadex 4.0 mg/kg (Vecuronium) (N=10) | Sugammadex 8.0 mg/kg (Vecuronium) (N=11)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Conjunctival irritation (Eye disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pupils unequal (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 | 3 (3) | 1 (1) | 1 (2) | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 3 (4) | 1 (1) | 3 (3) | 3 (3)
Chills (General disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Pain (General disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 0 | 1 (1) | 2 (2) | 0 | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 1 (1) | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0
Neuromuscular block prolonged (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0
Post procedural headache (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 2 (2) | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 | 1 (2) | 2 (2) | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 4 (5) | 2 (2) | 4 (4) | 3 (4) | 0 | 3 (3) | 3 (3) | 3 (4) | 3 (3)
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0/10
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Beta 2 microglobulin increased (Investigations) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0/10
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Headache (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 (3) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Haemorrhage (Vascular disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning the clinical trial described in the protocol will first be submitted to Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.